CLINICAL TRIAL: NCT06657586
Title: Investigation of the Effectiveness of Neuromuscular Exercise Program Accompanied by a Physiotherapist in Individuals With Degenerative Meniscal Tear
Brief Title: Investigation of the Effectiveness of Neuromuscular Exercise Program Accompanied With Degenerative Meniscal Tear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, hazal genc, Principal Investigator, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-10840098-202.3.02-3750
Record Dates: First submitted 2024-10-23; First posted 2024-10-24 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Meniscus Tear; Knee Injuries
Keywords: knee
MeSH Terms: conditions — Knee Injuries | interventions — Conservative Treatment

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- neuromuscular exercises (Experimental): Patients in group 1 received conservative treatment and neuromuscular exercises performed by a physiotherapist.
  Interventions: Other: neuromuscular exercises
- conservative treatment (Active Comparator): Patients in group 2 received conservative treatment
  Interventions: Other: conservative treatment

INTERVENTIONS:
Other: neuromuscular exercises — The exercise was applied in 18 sessions of 6 weeks.The treatment program included coldpack from cold application agent, ultrasound (US) treatment and TENS application from electrotherapy methods.
  Arms: neuromuscular exercises
Other: conservative treatment — The treatment program included coldpack from cold application agent, ultrasound (US) treatment and TENS application from electrotherapy methods.
  Arms: conservative treatment

SUMMARY:
The aim of the study was to investigate the effect of exercise program added to the treatment on physical function, postural balance, muscle strength, pain and gait in individuals with meniscal damage.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20-65 years.
* Having a meniscus tear.
* Volunteering to participate in the study.

Exclusion Criteria:

* Being diagnosed with a psychiatric illness.
* Having a neurological disease that may interfere with treatment.
* Having undergone meniscal surgery before.
* Having received physical therapy in the knee area in the last 6 months.
* Benefiting from any other treatment during the study.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2025-01-20 (Actual)

PRIMARY OUTCOMES:
Vertical jump | 6 weeks
  My Jump Lab 3 is a mobile application that precisely measures and analyzes vertical jump performance. It is an important tool to assess lower limb function and optimize treatment processes for patients with knee problems. The app provides key performance metrics such as jump height, flight time and strength and helps monitor patients' progress.
Star Balance Test | 6 weeks
  It is a test that evaluates dynamic balance and lower limb stability. The subject stands on one foot on eight radial lines drawn on the ground and tries to reach the farthest point of each line with the free foot. Reach distances in each direction are recorded and analyzed. This test is used to determine the risk of injury in athletes and to monitor balance development during rehabilitation.
Tegner Activity Level Scale | 6 weeks
  The Tegner Activity Level Scale is used to determine individuals' physical activity and level of sporting participation. The scale uses a scale ranging from 0 (sedentary) to 10 (professional athlete). This scale is particularly useful in the rehabilitation of sports injuries and for monitoring individuals' activity levels
KOOS-PS (Knee Injury and Osteoarthritis Outcome Score - Physical Function Short Form) | 6 weeks
  The KOOS-PS is used to assess the physiological and functional effects of knee osteoarthritis and knee injuries. The KOOS-PS includes five different knee-related subscales: Pain, Symptoms, Activities of Daily Living, Sports and Recreation, and Quality of Life. The physical function short form (PS) specifically assesses the impact of physical function on activities of daily living.
WOMET (Western Ontario Meniscal Evaluation Tool) | 6 weeks
  The WOMET is a specific scale developed to assess the symptoms and effects of meniscal injuries. It measures the pain, functional limitations, and impact on quality of life that patients experience with meniscal injuries.

CONTACTS AND LOCATIONS:
Locations (1):
- Bahçehir University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No